CLINICAL TRIAL: NCT05539885
Title: Optimal Timing of Parasternal Intercostal Nerve Block in Pediatric Patients Undergoing Cardiac Surgery
Brief Title: Parasternal Block in Pediatric Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ali Ahmed, Consultant of Anesthesia & Pain management, Faculty of Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Parasternal block
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pectointercostal Fascial Plane Block
Keywords: pectointercostal fascial plane block; pediatrics; open cardiac surgery; optimal timing
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-incisional PIFB (Active Comparator): Group P (ultrasound guided parasternal; PIFP block): patients will be injected with 0.4 mL/kg 0.25 bupivacaine in the fascial plane between the pectoralis major and internal intercostal muscles on each side of the sternum after induction of anesthesia and before skin incision under ultrasound guidance.
  Interventions: Procedure: Pre-incisional Ultrasound guided (PIFP) block
- Post-incisional PIFB (Active Comparator): Group S: After sternal closure, the surgeon will inject bupivacaine (0.5- to 2-mL aliquots depending on the weight) in the fascial plane under direct vision between the 5 anterior (2nd-6th) intercostal spaces on each side 1 to 1.5 cm lateral to the sternal edge using 25-gauge, 50 mm needle. The surgeon will inject the same dose and concentration of bupivacaine used in the ultrasound technique. This technique was prescribed before by Chaudhary et al (23).
  In both techniques, the maximum dose of bupivacaine will never be exceeded (2 mg/kg). In addition, all patients were administered 2 mL of 0.25% bupivacaine at the site of the mediastinal drain location.
  Interventions: Procedure: Post-incisional Surgeon delivered parasternal block group

INTERVENTIONS:
Procedure: Pre-incisional Ultrasound guided (PIFP) block — Patients in group P will be injected with 0.4 mL/kg of 0.25 bupivacaine in the fascial plane between the internal intercostal and pectoralis major muscles on each side of the sternum after induction of anesthesia and before skin incision under ultrasound guidance.
  Other Names: Pectointercostal fascial plane block
  Arms: Pre-incisional PIFB
Procedure: Post-incisional Surgeon delivered parasternal block group — After sternal closure, the surgeon will inject bupivacaine (0.5- to 2-mL aliquots depending on the weight) in the fascial plane under direct vision between the 5 anterior (2nd-6th) intercostal spaces on each side 1 to 1.5 cm lateral to the sternal edge using 25-gauge, 50 mm needle. The surgeon will inject the same dose and concentration of bupivacaine used in the ultrasound technique. This technique was prescribed before by Chaudhary et al (23).
  In both techniques, the maximum dose of bupivacaine will never be exceeded (2 mg/kg). In addition, all patients were administered 2 mL of 0.25% bupivacaine at the site of the mediastinal drain location.
  Arms: Post-incisional PIFB

SUMMARY:
The objective of this study is to determine whether the use of post-incisional surgeon-delivered parasternal block in children undergoing congenital heart surgery is associated with differences in outcomes when compared to ultrasound-guided pre-incisional parasternal block in the form of Pectointercostal fascial plane block (PIFB).

DETAILED DESCRIPTION:
Although many studies have found that pre-incisional parasternal block is effective in preventing postoperative sternotomy pain, we found no randomized controlled trials comparing pre-incisional vs post-incisional parasternal block in pediatric patients except for one retrospective cohort study done by Lisa et al comparing surgeon-delivered local anesthetic wound infiltration vs postoperative bilateral Petco-Intercostal Fascial Blocks. The post-incisional parasternal block may give prolonged postoperative pain control (equivalent to analgesia duration of pre-incisional parasternal block plus the duration of the operative procedure.)

ELIGIBILITY:
Inclusion Criteria:

Acyanotic Congenital heart disease; ASD (atrial septal defect), VSD (ventricular septal defect), and CAVC (common atrioventricular canal).

Elective open-heart surgery via median sternotomy and under CPB (cardiopulmonary bypass).

Hemodynamic stability (no evidence of heart failure, not on vasoactive drugs, and not on mechanical ventilation.

Exclusion Criteria:

Previous, urgent, or emergent cardiac surgery. Children with cyanotic congenital heart disease. local infection of the skin at the site of needle puncture, Allergy to bupivacaine, Coagulation disorders, Clinically significant liver or kidney disease, Heart failure or severe pulmonary hypertension.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesia request. | 24 hours
  The first analgesic request after extubation
Amount of rescue analgesia. | 24 hours
  Amount of rescue analgesia (total dose of fentanyl) after extubation.

SECONDARY OUTCOMES:
Postoperative pain score: | at extubation, 2nd, 6th, 12th, 16th, 20th, and 24th hour after extubation.
  Postoperative pain will be assessed by modified objective pain score (MOPS) in children at 0, 2, 6, 12, 16, 20, and 24 h after extubation. Wilson and Doyle modified the objective pain score by replacing blood pressure with posture. MOPS consists of 5 items (crying, movements, agitations, posture, and verbal). The minimum score is 0 (No pain) and the maximum is 10 (most sever pain).
Intraoperative fentanyl consumption | time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed Ali Ahmed, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollak U, Serraf A. Pediatric Cardiac Surgery and Pain Management: After 40 Years in the Desert, Have We Reached the Promised Land? World J Pediatr Congenit Heart Surg. 2018 May;9(3):315-325. doi: 10.1177/2150135118755977. PMID 29692232
- [Background] Roy N, Parra MF, Brown ML, Sleeper LA, Nathan M, Sefton BA, Baird CW, Mistry KP, Del Nido PJ. Initial experience introducing an enhanced recovery program in congenital cardiac surgery. J Thorac Cardiovasc Surg. 2020 Nov;160(5):1313-1321.e5. doi: 10.1016/j.jtcvs.2019.10.049. Epub 2019 Oct 24. PMID 31859070
- [Background] Zhang Y, Chen S, Gong H, Zhan B. Efficacy of Bilateral Transversus Thoracis Muscle Plane Block in Pediatric Patients Undergoing Open Cardiac Surgery. J Cardiothorac Vasc Anesth. 2020 Sep;34(9):2430-2434. doi: 10.1053/j.jvca.2020.02.005. Epub 2020 Feb 11. PMID 32151511